CLINICAL TRIAL: NCT00368823
Title: A Randomized Clinical Trial to Improve Prescribing Patterns in Ambulatory Pediatrics
Brief Title: A Trial of Point of Care Information in Ambulatory Pediatrics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HS10516-03
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2006-08-29 (Estimated); Status verified 2006-08

CONDITIONS: Acute Otitis Media; Allergic Rhinitis; Sinusitis; Constipation; Pharyngitis; Croup; Urticaria; Bronchiolitis
Keywords: point of care; evidence based medicine
MeSH Terms: conditions — Otitis Media; Rhinitis, Allergic; Sinusitis; Constipation; Pharyngitis; Croup; Urticaria; Bronchiolitis

INTERVENTIONS:
Device: Electronic point-of-care delivery system

SUMMARY:
Does presentation of clinical evidence for decision making at point-of-care improve prescribing patterns in ambulatory pediatrics?

DETAILED DESCRIPTION:
We showed previously that an electronic prescription writer and decision support system improved pediatric prescribing behavior for otitis media in an academic clinic setting. This study assessed whether point-of-care evidence delivery could demonstrate similar effects for a wide range of other common pediatric conditions. We performed a randomized controlled trial in a teaching clinic/clinical practice site and a primary care pediatric clinic serving a rural and semi-urban patient mix. There were 36 providers at the teaching clinic/practice site, and 8 providers at the private primary pediatric clinic, and an evidence-based message system presented real time evidence to providers based on prescribing practices for acute otitis media, allergic rhinitis, sinusitis, constipation, pharyngitis, croup, urticaria, and bronchiolitis. We measured the proportion of prescriptions dispensed in accordance with evidence.

ELIGIBILITY:
Inclusion Criteria: The 44 clinical providers at the two participating clinics. -

Exclusion Criteria: Study investigators

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44
Dates: Start 1999-11; Study Completion 2003-12

PRIMARY OUTCOMES:
prescribing practices for acute otitis media,
allergic rhinitis,
sinusitis,
constipation,
pharyngitis,
croup,
urticaria,
bronchiolitis

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Davis, MD, MPH, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Roosevelt Pediatric Clinic, Seattle, Washington
  - Skagit Valley Pediatrics, Skagit Valley, Washington